CLINICAL TRIAL: NCT01331122
Title: A Phase II, Double-Blind, Placebo-Controlled Randomized Crossover Study to Assess the Clinical Benefit and Safety of Droxidopa in the Treatment of Freezing of Gait Symptoms in Patients With Parkinson's Disease
Brief Title: Study to Assess Droxidopa in the Treatment of Freezing Of Gait Symptoms in Patients With Parkinson's Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Never initiated. Withdrawn by sponsor.
Sponsor: Chelsea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Droxidopa FOG201
Record Dates: First submitted 2010-10-13; First posted 2011-04-07 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Gait Disorders, Neurologic
MeSH Terms: conditions — Gait Disorders, Neurologic | interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- droxidopa (Experimental): Northera (2R,3S)-2-amino-3-(3,4-dihydroxyphenyl)-3-hydroxypropanoic acid L-DOPS L-threo-dihydroxyphenylserine Droxidopa SM-5688
  Interventions: Drug: droxidopa
- placebo (Placebo Comparator): placebo
  Interventions: Drug: droxidopa

INTERVENTIONS:
Drug: droxidopa — Oral, 100, 200, 300, 400, 500, or 600 mg TID, duration includes two crossover periods of up to a 2 week titration period followed by a 4 week treatment period,with a washout between crossover periods.
  Other Names: Northera; SM-5688; L-DOPS; L-threo-dihydroxyphenylserine

SUMMARY:
Freezing of Gait (FoG) is a class of symptoms that occur in Parkinson's patients. Also called motor blocks, FoG is characterized by a sudden inability to move the lower extremities which usually lasts less than 10 seconds. The exact pathophysiology of FoG is poorly understood, but treatment with levodopa appears to improve FoG observed in the off-state. As Parkinson's patients progress in severity, FoG in the on-state can increase in frequency and appears to be resistant to dopaminergic therapies. There is additional evidence that norepinephrine as well as dopaminergic systems may be involved in FoG.

Droxidopa has has been approved for use in Japan since 1989 for treatment of frozen gait or dizziness associated with Parkinson's Disease. This study is to further explore the safety and efficacy of droxidopa in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged at least 30 years;
* Diagnosed with probable levodopa-responsive idiopathic Parkinson's Disease , and receiving levodopa. Other Parkinson's Disease medications can also be used.
* At least 3 months incidence of typical freezing of gait (FOG) symptoms, occurring while levodopa is otherwise providing an "on" mobility state (including at least one of the following FOG patterns: start hesitancy, freezing at making turns or when passing through a doorway, spontaneous freezing during continued walking, or freezing of gait related to a simultaneous mental or physical activity).
* Provide written informed consent to participate in the study and understand that they may withdraw their consent at any time without prejudice to their future medical care
* On a stable dose of carbidopa, alone or with other Parkinson's medication, providing a range of carbidopa between 100mg and 400mg daily

Exclusion Criteria:

* Taking direct acting vasoconstricting agent (i.e. ephedrine or midodrine). Patients taking vasoconstrictor agents such as ephedrine or midodrine must stop taking these drugs at least 2 days or 5 half-lives (whichever is longer) prior to their baseline visit;
* Taking more than one anti-hypertensive medication for the treatment of high blood pressure. Short acting anti-hypertensive medication taken at night to prevent supine hypertension will be allowed.
* Have changed dose or frequency of Parkinson's medication within 2 weeks of baseline
* Known or suspected alcohol or substance abuse within 1 year
* Sustained hypertension (BP greater than 140/90 mmHg in the sitting position)
* Symptomatic coronary artery disease, severe congestive heart failure
* Women who are pregnant, lactating, or plan to become pregnant during the course of this study;
* Women of child bearing potential (WOCP) who are not using two methods of contraception (at least one barrier: i.e. condom) with their partner.
* Male patients who are sexually active with a woman of child bearing potential (WOCP) and not using two methods of contraception (at least one barrier: i.e. condom)
* Untreated closed angle glaucoma, or treated closed angle glaucoma that in the opinion of an ophthalmologist would cause increased risk to the patient;
* Active (last 6 months) atrial fibrillation or, in the investigator's opinion, any other significant cardiac arrhythmia that should preclude the patient from this trial;
* History of myocardial infarction or unstable angina
* Diabetes insipidus, insulin dependent diabetes mellitus, or diabetic neuropathy;
* In the investigator's opinion, any other significant systemic illness;
* Known or suspected malignancy (other than basal cell carcinoma);
* Known gastrointestinal illness or other gastrointestinal disorder that may, in the investigator's opinion, affect the absorption of study drug;
* Any major surgical procedure within 30 days of the baseline visit;
* Currently receiving any investigational drug or have received an investigational drug within 30 days of the baseline visit;
* In the investigator's opinion, clinically significant abnormalities on clinical examination or laboratory testing that should preclude the patient from this trial;
* Patient has only lower body Parkinson's Disease
* In the investigators opinion, freezing of gait is attributable to previous stroke

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of droxidopa as measured by the incidence, relatedness, and severity of adverse events. | 18 Weeks

SECONDARY OUTCOMES:
Evaluate the effect of droxidopa on freezing of gait symptoms using the Freezing of Gait Questionnaire | 18 Weeks
Evaluate the efficacy of droxidopa in the treatment of freezing of gait by using the Observed Freezing of Gait Rating (OFGR) scale | 18 Weeks
Evaluate the effect of droxidopa on signs and symptoms associated with Parkinson's Disease utilizing the composite scores of the Unified Parkinson's Disease Rating Scale | 18 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter A LeWitt, MD, Principal Investigator — Henry Ford Hospital
Locations (2):
- Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan, United States
- University of Alberta, Movement Disorders Clinic Glenrose Rehabilitation Hospital, Edmonton, Alberta, Canada